CLINICAL TRIAL: NCT03835286
Title: Vitamin C to Reduce Exogenous Vasopressor Dose in Septic Shock; a Randomized Clinical Trial
Brief Title: Vitamin C to Reduce Vasopressor Dose in Septic Shock
Acronym: ViCiS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: COVID 19
Sponsor: Hospital Español de Mexico (Other)
Responsible Party: Principal Investigator, Jose J Zaragoza, MD, Clinical Professor, Hospital Español de Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EHE0042
Record Dates: First submitted 2019-01-22; First posted 2019-02-08 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Septic Shock; Sepsis
Keywords: critical care; vitamin C; vasopressor; intensive care unit
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C (Experimental): Vitamin C experimental group
  Interventions: Drug: Vitamin C
- Control (Placebo Comparator): Placebos Controlled group
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Vitamin C — 6 grams of Vitamin C in 250 ml of 0.9% saline in continuous infusion for 24 hours, 3 doses.
  Other Names: Ascorbic Acid
  Arms: Vitamin C
Drug: Placebos — Placebos: 250 ml of 0.9% saline in continuous infusion for 24 hours, 3 doses.
  Other Names: Placebo
  Arms: Control

SUMMARY:
Randomized, controlled, double blind clinical trial. Adult patients admitted to the ICU of the Hospital Español de México with a diagnosis of septic shock will be included.

Patients will be randomized to one of the study groups:

Intervention Group: Vitamin C 6 grams in 250 ml of 0.9% saline solution every 24 hours, in continuous infusion for 72 hours.

Placebo Group: 0.9% saline solution 250 ml every 24 hours, in continuous infusion for 72 hours.

DETAILED DESCRIPTION:
Randomized, controlled, double blind clinical trial. Adult patients admitted to the ICU of the Hospital Español de México with a diagnosis of septic shock will be included.

Patients will be randomized to one of the study groups:

Intervention Group: Vitamin C 6 grams in 250 ml of 0.9% saline solution every 24 hours, in continuous infusion for 72 hours.

Placebo Group: 0.9% saline solution 250 ml every 24 hours, in continuous infusion for 72 hours.

Bottles will be identical, only identified by the sequential number of the patient that has been included.

Primary objective is to demonstrate that the administration of intravenous Vitamin C decreases the dose of exogenous vasopressors in patients with septic shock

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Septic Shock

Exclusion Criteria:

* Previous treatment exceeded 24 hours
* Refusal to participate
* Do Not Resuscitate
* Participation in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Vasopressor dose | 72 hours
  Hourly dose of exogenous vasopressor

SECONDARY OUTCOMES:
Hours of vasopressor use | through study completion, an average of 30 days
  Total hours of vasopressor use
Days of mechanical ventilation | through study completion, an average of 30 days
  Total days of mechanical ventilation use
Days of Intensive Care Unit stay | through study completion, an average of 30 days
  Total days of intensive care unit stay
Mortality in Intensive Care Unit | through study completion, an average of 30 days
  Rate of intensive care mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo Martinez-Zubieta, MD, Study Chair — Hospital Español de Mexico
Locations (1):
- Hospital Español, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Complete database will be shared as requested by the publishing journal, once the study is completed
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Available one year after
Access Criteria: Journal provided